CLINICAL TRIAL: NCT04230161
Title: Estimating the Malaria Prevention Impact of New Nets: Observational Analyses to Evaluate the Evidence Generated During Piloted New Net Distributions in Rwanda
Status: Completed | Type: Observational
Sponsor: PATH (Other)
Collaborators: Rwanda Biomedical Centre (Other); University of Rwanda (Other); Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 1409734-2
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Malaria
Keywords: Long-lasting insecticidal net; LLIN; Insecticide treated net; ITN; Malaria; Epidemiology; Anthropology; Durability; Cost-effectiveness
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Standard LLIN: This group receives Yahe LN ITNs during the mass distribution campaign.
  Interventions: Other: Standard long-lasting insecticidal net
- Chlorfenapyr ITN: This group receives Interceptor G2 ITNs during the mass distribution campaign.
  Interventions: Other: Chlorfenapyr insecticide treated net
- Standard LLIN and IRS: This group receives Yahe LN ITNs during the mass distribution campaign and IRS.
  Interventions: Other: Standard long-lasting insecticidal net; Other: Indoor residual spraying

INTERVENTIONS:
Other: Standard long-lasting insecticidal net — Yahe LN (Yamei Industry) contains a pyrethroid insecticide.
  Other Names: Yahe LN
  Groups: Standard LLIN; Standard LLIN and IRS
Other: Chlorfenapyr insecticide treated net — Interceptor G2® (BASF) is an ITN containing two active ingredients: Alpha-cypermethrin, a pyrethroid insecticide, and chlorfenapyr, a pyrrole insecticide.
  Other Names: Interceptor G2®
  Groups: Chlorfenapyr ITN
Other: Indoor residual spraying — Fludora Fusion (Bayer Vector Control) is a spray containing two active ingredients: clothianidin, a neonicotinoid insecticide, and deltamethrin, a pyrethroid insecticide.
  Other Names: Fludora Fusion
  Groups: Standard LLIN and IRS

SUMMARY:
The use of insecticide-treated bed nets (ITNs) has contributed to the substantial reduction in malaria cases and deaths. This progress is threatened by increasing resistance in mosquito populations to commonly used insecticides. Newly developed, next-generation ITNs using two insecticides or an insecticide synergist and an insecticide are effective against resistant mosquitoes, but large-scale uptake of these nets has been slow due to higher costs and lack of enough evidence to support broad policy recommendations.

This observational study will occur alongside a pilot distribution of next-generation ITNs and collect data over three years on their entomological and epidemiological impact as well as anthropological factors that influence their uptake and use. Enhanced data collection will occur in three districts: one district that will receive Interceptor G2 ® ITN (BASF) and two comparator districts, one that will receive standard pyrethroid-only ITNs and one that will receive standard pyrethroid-only ITNs and indoor residual spraying (IRS). Data will be collected on malaria vector bionomics, disease epidemiology, and human behaviors in order to help better demonstrate the public health value of next-generation ITNs and to support donors, policymakers, and National Malaria Control Programs in their ITN decision-making and planning processes.

DETAILED DESCRIPTION:
The World Health Organization's (WHO) 2018 World Malaria Report estimates that in 2017, 219 million cases of malaria occurred worldwide resulting in 435,000 deaths, 93% of which occurred in Africa (WHO 2018). While this represents a remarkable improvement in comparison with 2000, with malaria deaths having fallen by 40% in Africa, the downward trends in incidence and mortality stalled between 2015 and 2017. This recent failure to maintain the hard-won progress, let alone accelerate progress towards elimination, over the past three years has caused WHO to describe the global fight against malaria as being at a cross roads, calling for increased funding and highlighting the need to develop, optimize, and implement new tools to combat malaria.

Universal coverage of populations at risk with malaria vector control interventions-primarily insecticide treated nets (ITNs) and indoor residual spraying (IRS)-in malaria-endemic countries is a global and national priority because of its fundamental importance for malaria control and elimination. Unfortunately, the effectiveness of these tools is threatened by the emergence and spread of pyrethroid resistance in key mosquito populations, which is now reported in more than 85% of all malaria-endemic countries and poses significant risk to the future impact of these tools. Emerging evidence suggests, however, that increasing mosquito mortality-and thereby continuing to reduce malaria transmission-is possible in areas with pyrethroid resistance by introducing new insecticide formulations for IRS and ITNs. For example, Protopopoff et al. showed in Tanzania that the distribution of LLINs with PBO plus pyrethroid reduced malaria prevalence by 13% compared to standard pyrethroid-only LLIN distribution (42% vs. 29%; p=0.0011), and Tiono et al., working in Burkina Faso, showed that the distribution of a dual active-ingredient ITN reduced clinical malaria incidence by 22% (Incidence Rate Ratio = 0.88; p=0.04) and potentially infective mosquito bites by 51% (entomological inoculation rate ratio = 0.49; p<0.0001) compared to the distribution of a standard pyrethroid-only LLIN.

While there is evidence that standard LLINs can continue to provide effective personal protection to regular net users in regions with resistant vector populations, new classes of ITNs developed to perform against pyrethroid-resistant mosquitoes have been developed, with early trials and modelling suggesting that they may provide superior protective efficacy against malaria in areas with pyrethroid-resistant vectors. Access to these new resistance-breaking ITNs is restricted by the need for efficacy data for continuing policy recommendations, high prices, lack of evidence of cost effectiveness compared to pyrethroid-only LLINs, and consequent poor demand in an uncertain market. Interceptor® G2 (IG2) (BASF), a new type of ITN consisting of two active ingredients including a mixture of a pyrethroid (alpha-cypermethrin) and a pyrrole (chlorfenapyr) insecticide, recently achieved WHO prequalification listing demonstrating that it performs to the thresholds required of pyrethroid-only LLINs and has no known specific side effects. While the IG2 ITN has been subsequently registered and approved for use in Rwanda based on this WHO listing, the Roll Back Malaria Vector Control Advisory Group guidance indicates that dual active ingredient ITNs will require further epidemiological evidence before policy recommendations are made for their use in preference to pyrethroid-only LLINs in certain settings.

The Global Fund and Unitaid have developed a market shaping project for IG2 and other ITNs with novel insecticide formulations. Evidence on the efficacy of IG2s will be generated by the project through two randomized control trials taking place in Benin and Tanzania. In addition, through this project, these next-generation ITNs will be made available to countries for incorporation into their national distribution programs as pilot distributions with the aim of determining real-world effectiveness and cost-effectiveness in different contexts. In addition to the pilot distribution of IG2s taking place in Rwanda, four other countries will be piloting IG2s as part of the New Nets Project: Burkina Faso, Mali, Mozambique, and Nigeria. This research will utilize these pilot distributions to understand the cost-effectiveness of the new ITNs in the chosen settings. The NMCP in Rwanda, in discussion with the Global Fund, chose to incorporate IG2 ITNs into the upcoming 2019 mass distribution campaign. This study will gather information to determine the public health impact of the IG2 ITNs in Rwanda, in comparison to sites that will receive standard pyrethroid-only LLINs or standard pyrethroid-only LLINs and IRS. The aim of this research is to better understand the effectiveness and cost effectiveness of IG2 ITNs in Rwanda and to collect data on community uptake of the ITNs. During the upcoming pilot implementation, entomological, epidemiological, and anthropological data will be collected in three study districts, one that will receive IG2 ITNs, one comparator district that will receive standard LLINs, and one additional comparator district that will receive standard LLINs with IRS. Data will be analyzed and results disseminated to support the NMCP, donors, policymakers, and other national and regional stakeholders in their ITN decision-making and planning processes. Each component specifically aims to:

* Epidemiological component - measure the epidemiological impact of the new IG2 ITNs and standard LLINs in real deployment scenarios through observational studies. These studies will compare trends in (1) malaria case incidence rates passively reported to the national health system (passive case detection, PCD) and (2) malaria infection prevalence, measured through Rapid Diagnostic Tests (RDTs), in participants 6 months of age and older from annual cross-sectional surveys during peak transmission periods.
* Entomological component - evaluate the impact of IG2 ITNs on vector populations and biting rates, compared to standard LLINs, through national mosquito surveillance data that will measure trends in species-specific (1) adult vector densities (2) indoor and outdoor human landing rates (3) estimated entomological inoculation rates and (4) insecticide resistance patterns.
* Anthropological component - map the social determinants of impact for IG2 LLINs and determine transmission risk defined as the intersection between time at risk of mosquito blood feeding and human activities not under protection of an ITNN, through gathering evidence on LLIN uptake and usage. The collection of reliable data using observation, focus group discussions, and key informant interviews is an essential component of the evaluation for both modeling and contextual analysis of impact.
* Costing and cost-effectiveness component - estimate the cost and cost-effectiveness of IG2 ITNs in Rwanda through data on the price of the product, delivery and deployment costs, and product effectiveness based on case incidence rates measured during the epidemiological component of this study. Additionally, mean costs per case averted that might occur in other contexts will be modeled and incorporated into the cost-effectiveness evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Passive data collection: all suspected malaria cases (fevers) that self-present to the national health system and are counted in the district health surveillance systems.
* Cross sectional survey: Households in the district.

  * Residents of the household visited.
  * Questionnaire: any adult member of the household .
  * Malaria screening: all members aged 6 months or older from the above consenting household.
* Individuals of box sexes, not belonging to vulnerable categories (those with cognitive impairment or other person for whom full and open consent cannot be guaranteed) (Key informant interviews, focus group discussions, and participant observations).
* Individuals 18 years old and above (Key informant interviews, focus group discussions, and observations).
* Individuals of both sexes regardless of age (observations).

Exclusion Criteria:

* District non-residents.
* Malaria screening: history of recent (within one month) malaria infection or treatment with anti-malarial medication (cross-sectional).
* Parents or guardians who have not yet reached age of consent (18 years) and their children will not be included in study activities requiring consent.
* Individuals belonging to vulnerable categories (key informant interviews, focus group discussions, observations).
* Individuals unwilling and/or unable of giving consent (key informant interviews, focus group discussions, observations).
* Individuals below age of consent (20 years) (key informant interviews, focus group discussions, observations).
* Heads of households unwilling and/or unable of giving consent (observations).
* Individuals who do not wish to be included in observations will be excluded (observations).

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Households selected for enrollment in the cross-sectional survey will be randomly selected from each of the three study districts: Ruhango, Nyamagabe, and Karongi. All members of the selected households will be asked to participate in the malaria biomarker survey to test for malaria using an RDT.
  The villages selected for anthropological surveillance will be the same as those used for entomological surveillance.
  Passive case detection data will include all malaria tests recorded in all health facilities in the three study districts.
Sampling Method: Probability Sample
Enrollment: 3502 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Cumulative malaria incidence | November 2019 to December 2022, monthly
  Malaria incidence measured through passive case detection at health facilities in each district. This measure accounts for symptomatic cases self-reporting to the formal health system for care.

SECONDARY OUTCOMES:
Vector species composition | December 2019 to December 2022, monthly
  All Anopheles mosquitoes sampled during Centers for Disease Control and Prevention light traps (CDCLT) and human landing collections (HLC) will be identified morphologically to species group
Species-specific population densities | December 2019 to December 2022, monthly
  Based on Anopheles mosquitoes sampled during CDCLT
Biting behaviors | December 2019 to December 2022, monthly
  Based on Anopheles mosquitoes sampled during CDCLT
Estimated entomological inoculation rates | December 2019 to December 2022, monthly
  Based on Anopheles mosquitoes sampled during CDCLT and HLC
Insecticide resistance profile | December 2019 to December 2022, monthly
  Measurement of kdr and ace-1 mutation frequencies, WHO tube bioassays at minimum and CDC bottle bioassays to characterize insecticide resistance intensity
Parasite prevalence in children 6 months or older | January 2020, January 2021, January 2022
  Prevalence calculated from cross-sectional surveys conducted during the peak transmission season

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Wagman, PhD, Principal Investigator — PATH; Aimable Mbituyumuremyi, MD, Principal Investigator — Rwanda Biomedical Centre
Locations (1):
- Rwanda Biomedical Centre, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alonso P, Noor AM. The global fight against malaria is at crossroads. Lancet. 2017 Dec 9;390(10112):2532-2534. doi: 10.1016/S0140-6736(17)33080-5. Epub 2017 Nov 29. No abstract available. PMID 29195688
- [Background] Bass C, Nikou D, Donnelly MJ, Williamson MS, Ranson H, Ball A, Vontas J, Field LM. Detection of knockdown resistance (kdr) mutations in Anopheles gambiae: a comparison of two new high-throughput assays with existing methods. Malar J. 2007 Aug 13;6:111. doi: 10.1186/1475-2875-6-111. PMID 17697325
- [Background] Bayili K, N'do S, Namountougou M, Sanou R, Ouattara A, Dabire RK, Ouedraogo AG, Malone D, Diabate A. Evaluation of efficacy of Interceptor(R) G2, a long-lasting insecticide net coated with a mixture of chlorfenapyr and alpha-cypermethrin, against pyrethroid resistant Anopheles gambiae s.l. in Burkina Faso. Malar J. 2017 May 8;16(1):190. doi: 10.1186/s12936-017-1846-4. PMID 28482891
- [Background] Bhatt S, Weiss DJ, Cameron E, Bisanzio D, Mappin B, Dalrymple U, Battle K, Moyes CL, Henry A, Eckhoff PA, Wenger EA, Briet O, Penny MA, Smith TA, Bennett A, Yukich J, Eisele TP, Griffin JT, Fergus CA, Lynch M, Lindgren F, Cohen JM, Murray CLJ, Smith DL, Hay SI, Cibulskis RE, Gething PW. The effect of malaria control on Plasmodium falciparum in Africa between 2000 and 2015. Nature. 2015 Oct 8;526(7572):207-211. doi: 10.1038/nature15535. Epub 2015 Sep 16. PMID 26375008
- [Background] Fornadel CM, Norris LC, Franco V, Norris DE. Unexpected anthropophily in the potential secondary malaria vectors Anopheles coustani s.l. and Anopheles squamosus in Macha, Zambia. Vector Borne Zoonotic Dis. 2011 Aug;11(8):1173-9. doi: 10.1089/vbz.2010.0082. Epub 2010 Dec 13. PMID 21142969
- [Background] Hakizimana E, Karema C, Munyakanage D, Githure J, Mazarati JB, Tongren JE, Takken W, Binagwaho A, Koenraadt CJM. Spatio-temporal distribution of mosquitoes and risk of malaria infection in Rwanda. Acta Trop. 2018 Jun;182:149-157. doi: 10.1016/j.actatropica.2018.02.012. Epub 2018 Feb 21. PMID 29476726
- [Background] Kleinschmidt I, Bradley J, Knox TB, Mnzava AP, Kafy HT, Mbogo C, Ismail BA, Bigoga JD, Adechoubou A, Raghavendra K, Cook J, Malik EM, Nkuni ZJ, Macdonald M, Bayoh N, Ochomo E, Fondjo E, Awono-Ambene HP, Etang J, Akogbeto M, Bhatt RM, Chourasia MK, Swain DK, Kinyari T, Subramaniam K, Massougbodji A, Oke-Sopoh M, Ogouyemi-Hounto A, Kouambeng C, Abdin MS, West P, Elmardi K, Cornelie S, Corbel V, Valecha N, Mathenge E, Kamau L, Lines J, Donnelly MJ. Implications of insecticide resistance for malaria vector control with long-lasting insecticidal nets: a WHO-coordinated, prospective, international, observational cohort study. Lancet Infect Dis. 2018 Jun;18(6):640-649. doi: 10.1016/S1473-3099(18)30172-5. Epub 2018 Apr 9. PMID 29650424
- [Background] Koekemoer LL, Kamau L, Hunt RH, Coetzee M. A cocktail polymerase chain reaction assay to identify members of the Anopheles funestus (Diptera: Culicidae) group. Am J Trop Med Hyg. 2002 Jun;66(6):804-11. doi: 10.4269/ajtmh.2002.66.804. PMID 12224596
- [Background] Protopopoff N, Mosha JF, Lukole E, Charlwood JD, Wright A, Mwalimu CD, Manjurano A, Mosha FW, Kisinza W, Kleinschmidt I, Rowland M. Effectiveness of a long-lasting piperonyl butoxide-treated insecticidal net and indoor residual spray interventions, separately and together, against malaria transmitted by pyrethroid-resistant mosquitoes: a cluster, randomised controlled, two-by-two factorial design trial. Lancet. 2018 Apr 21;391(10130):1577-1588. doi: 10.1016/S0140-6736(18)30427-6. Epub 2018 Apr 11. PMID 29655496
- [Background] Ranson H, N'guessan R, Lines J, Moiroux N, Nkuni Z, Corbel V. Pyrethroid resistance in African anopheline mosquitoes: what are the implications for malaria control? Trends Parasitol. 2011 Feb;27(2):91-8. doi: 10.1016/j.pt.2010.08.004. Epub 2010 Sep 16. PMID 20843745
- [Background] Scott JA, Brogdon WG, Collins FH. Identification of single specimens of the Anopheles gambiae complex by the polymerase chain reaction. Am J Trop Med Hyg. 1993 Oct;49(4):520-9. doi: 10.4269/ajtmh.1993.49.520. PMID 8214283
- [Background] Sherrard-Smith E, Griffin JT, Winskill P, Corbel V, Pennetier C, Djenontin A, Moore S, Richardson JH, Muller P, Edi C, Protopopoff N, Oxborough R, Agossa F, N'Guessan R, Rowland M, Churcher TS. Systematic review of indoor residual spray efficacy and effectiveness against Plasmodium falciparum in Africa. Nat Commun. 2018 Nov 26;9(1):4982. doi: 10.1038/s41467-018-07357-w. PMID 30478327
- [Background] Tiono AB, Ouedraogo A, Ouattara D, Bougouma EC, Coulibaly S, Diarra A, Faragher B, Guelbeogo MW, Grisales N, Ouedraogo IN, Ouedraogo ZA, Pinder M, Sanon S, Smith T, Vanobberghen F, Sagnon N, Ranson H, Lindsay SW. Efficacy of Olyset Duo, a bednet containing pyriproxyfen and permethrin, versus a permethrin-only net against clinical malaria in an area with highly pyrethroid-resistant vectors in rural Burkina Faso: a cluster-randomised controlled trial. Lancet. 2018 Aug 18;392(10147):569-580. doi: 10.1016/S0140-6736(18)31711-2. Epub 2018 Aug 10. PMID 30104047
- [Background] Weill M, Malcolm C, Chandre F, Mogensen K, Berthomieu A, Marquine M, Raymond M. The unique mutation in ace-1 giving high insecticide resistance is easily detectable in mosquito vectors. Insect Mol Biol. 2004 Feb;13(1):1-7. doi: 10.1111/j.1365-2583.2004.00452.x. PMID 14728661
- See also: Bernard, HR. Research Methods in Anthropology: Qualitative and Quantitative Approaches. 4th — http://www.dphu.org/uploads/attachements/books/books_476_0.pdf
- See also: Ben-Shlomo Y, Brookes S, Hickman M. Lecture Notes: Epidemiology, Evidence-based Medicine and Public Health. — https://www.wiley.com/en-us/Lecture+Notes%3A+Epidemiology%2C+Evidence+based+Medicine+and+Public+Health%2C+6th+Edition-p-9781444334784
- See also: Malaria and Other Parasitic Diseases Division (MOPDD) of the Rwanda Biomedical Center Ministry of Health. National Guidelines for the Treatment of Malaria in Rwanda. — http://elearning.moh.gov.rw/pluginfile.php/3000/course/overviewfiles/National%20Guidelines%20for%20the%20Treatment%20of%20Malaria%20in%20Rwanda.pdf
- See also: Malaria and Other Parasitic Diseases Division (MOPDD) of the Rwanda Biomedical Center Ministry of Health and ICF. Rwanda Malaria Indicator Survey (RMIS) 2017 — https://www.dhsprogram.com/pubs/pdf/MIS30/MIS30.pdf
- See also: National Institute of Statistics of Rwanda (NISR), Ministry of Health (MOH) [Rwanda], and ICF International. Rwanda Demographic and Health Survey 2014 - 15 — https://dhsprogram.com/pubs/pdf/FR316/FR316.pdf
- See also: The US President's Malaria Initiative (PMI) Africa Indoor Residual Spraying (AIRS) Project. The PMI AIRS Project Semi-Annual Report: October 1, 2016 - March 31, 2017. — https://www.pmi.gov/docs/default-source/default-document-library/implementing-partner-reports/africa-indoor-residual-spraying-project-semi-annual-report-(october-2016---march-2017).pdf
- See also: The US President's Malaria Initiative (PMI). Rwanda: Malaria Operational Plan FY 2019. — https://www.pmi.gov/docs/default-source/default-document-library/malaria-operational-plans/fy19/fy-2019-rwanda-malaria-operational-plan.pdf
- See also: United Nations (UN). Outreach Programme on the Rwanda Genoicde and the United Nations. — https://www.un.org/en/preventgenocide/rwanda/
- See also: Malkki, L., 1995. Purity and Exile: Violence, Memory, and National Cosmology. — https://www.press.uchicago.edu/ucp/books/book/chicago/P/bo3624883.html
- See also: Lévi-Strauss, C., 1969. The elementary structures of kinship (No. 340). — https://www.worldcat.org/title/elementary-structures-of-kinship/oclc/720027839